CLINICAL TRIAL: NCT01395082
Title: ACAM2000® Myopericarditis Registry
Status: Completed | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: H-406-003; U1111-1120-1721 (Other: WHO)
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Myocarditis; Pericarditis
Keywords: Myocarditis; Pericarditis; Vaccinia virus; ACAM2000®; Smallpox vaccine
MeSH Terms: conditions — Myocarditis; Pericarditis; Vaccinia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Entire registry group: Participants with potential myopericarditis cases referred to the Registry

SUMMARY:
The purpose of this registry is to study the natural history of vaccination-related myocarditis and pericarditis and to assess possible risk factors for these conditions.

Primary Objective:

- To document the natural history of confirmed, probable, suspected, and subclinical myocarditis and pericarditis (myopericarditis) following ACAM2000® vaccination.

Other Pre-defined Objective:

- To look for potential predictive factors for the prognosis of myopericarditis following ACAM2000® vaccination.

DETAILED DESCRIPTION:
All participants will have received previous vaccination with ACAM2000 but will not receive any vaccination as part of the registry. All participants enrolled in the registry will be followed for 2 up to 5 years (depending on whether there are persisting signs and symptoms of myopericarditis).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are current or former members of the active duty, Reserve, or National Guard, from any branch of service
* Documented vaccination with ACAM2000® vaccine
* Meet one of the case definitions for suspect, probable, confirmed or subclinical myopericarditis.

Exclusion Criteria:

* Individuals not meeting at least one of the case definitions for myopericarditis will not be entered into the Registry.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants will have received previous vaccination with ACAM2000® but will not receive any vaccination as part of the registry.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
The number of confirmed, probable, suspected, and subclinical cases of myopericarditis, categorized by time since vaccination | 2 years after enrollment or after the last symptoms or positive findings

OTHER OUTCOMES:
The natural history of myopericarditis in terms of time to resolution or change in status of myopericarditis and the pattern of changes in status of myopericarditis | 2 years after enrollment or after the last symptoms or positive findings

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Emergent BioSolutions
Locations (1):
- San Diego, California, United States